CLINICAL TRIAL: NCT01719159
Title: Intrathecal Therapy With Monoclonal Antibodies in Progressive Multiple Sclerosis
Acronym: ITT-PMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Svenningsson (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Sponsor-Investigator, Anders Svenningsson, MD, PhD, Assoc Prof, Umeå University
Organization: Umeå University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITT-PMS
Record Dates: First submitted 2012-10-25; First posted 2012-11-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Progressive multiple sclerosis; Monoclonal antibodies; Mabthera; Intrathecal treatment
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): Rituximab, 25 mg, is administrated intrathecal three times one week apart
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 25 mg rituximab is injected intrathecally via an Ommaya reservoir once a week for 3 weeks. Patients are then followed for one year.
  Other Names: Mabthera

SUMMARY:
This is a is a small scale open phase two interventional study to assess long-term stabilising effects of on neurological symptoms by regular intrathecal administered monoclonal antibodies in progressive multiple sclerosis.

DETAILED DESCRIPTION:
There is presently no efficient therapy available in progressive MS, especially if there is no clear evidence of active inflammatory lesions or exacerbations as part of the disease. There are, however, evidence that some treatment protocols using cytotoxic drugs may to some extent slow down the progressive course. One specific feature of long-standing MS is that inflammatory cells accumulate in the central nervous system(CNS) compartment in the subarachnoid and perivascular spaces and may therefore be hard to reach via standard drug delivery through systemic administration. Administration of substances via the Intrathecal (IT) route, however, have shown to efficiently distribute in the subarachnoid spaces and may therefore be an attractive route of drug delivery

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 and 65 years of age (nonfertile women or fertile women with effective contraceptive methods)
* Progressive MS since at least three years
* Some kind of documented progression of neurological symptoms during the previous two years.
* Expanded Disability Status Scale (EDSS) 4,0 - 7.0 (inclusive) (basically spared arm functions)
* Conventional therapy not indicated, contraindicated or failed
* Judged as compliant with the protocol

Exclusion Criteria:

* Eligible for any of the conventional MS therapies
* Relapsing remitting multiple sclerosis (RRMS)
* Bleeding diathesis or medication contraindicating neurosurgical procedures or lumbar puncture
* Cognitive defect making informed consent unreliable
* Any medical condition contraindicating minor surgical procedures, as judged by anaesthesiologist
* Severe, uncontrolled heart disease
* Pregnant or lactating women
* Patients having contraindication for or otherwise not compliant with MRI investigations
* Documented vulnerability to infections
* Simultaneous treatment with other immunosuppressive drugs
* Documented allergy or intolerance to Rituximab
* Severe psychiatric condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | One year after completed treatment
  Feasibility of IT administered monoclonal antibodies

SECONDARY OUTCOMES:
Stabilisation of the neurological deterioration | At 3,6,9,12 month after completed treatment
  Questionaires regarding MS quality of life, symptom inventory and fatigue will be used.

OTHER OUTCOMES:
Immunological markers in blood | At 3,6,9,12 month after treatment
  I.e. absolute numbers of major lymphocyte subset as well as regulatory cell subset
Immunological markers in cerebrospinal fluid (CSF) | At 3, 6, 9 12 month after treatment
  I.e. absolute numbers of major lymphocyte subset as well as regulatory cell subset

CONTACTS AND LOCATIONS:
Overall Officials: Anders Svenningsson, MD, PhD, Principal Investigator — Umea university
Locations (2):
- Sweden (2):
  - Department of neurology, Umeå University Hospital, Umeå
  - Dept of neurology, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request from the researcher or scientific journals

REFERENCES:
- [Derived] Bergman J, Burman J, Gilthorpe JD, Zetterberg H, Jiltsova E, Bergenheim T, Svenningsson A. Intrathecal treatment trial of rituximab in progressive MS: An open-label phase 1b study. Neurology. 2018 Nov 13;91(20):e1893-e1901. doi: 10.1212/WNL.0000000000006500. Epub 2018 Oct 10. PMID 30305449
- [Derived] Bergman J, Dring A, Zetterberg H, Blennow K, Norgren N, Gilthorpe J, Bergenheim T, Svenningsson A. Neurofilament light in CSF and serum is a sensitive marker for axonal white matter injury in MS. Neurol Neuroimmunol Neuroinflamm. 2016 Aug 2;3(5):e271. doi: 10.1212/NXI.0000000000000271. eCollection 2016 Oct. PMID 27536708